CLINICAL TRIAL: NCT06593600
Title: A Phase 2 Double-Blind Placebo-Controlled Single-Dose Study of Pharmacodynamics, Pharmacokinetics, Safety, and Tolerability of REGN7544, an NPR1 Antagonist Monoclonal Antibody, in Patients With Postural Orthostatic Tachycardia Syndrome
Brief Title: Study of Natriuretic Peptide Receptor 1 (NPR1) Antagonist in Adult Patients With Postural Orthostatic Tachycardia Syndrome (POTS)
Acronym: PINNACLE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R7544-POTS-2429
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS)
Keywords: Orthostatic intolerance
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Randomized 1:1:1
  Interventions: Drug: REGN7544
- High Dose (Experimental): Randomized 1:1:1
  Interventions: Drug: REGN7544
- Matching Placebo (Placebo Comparator): Randomized 1:1:1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN7544 — Subcutaneous (SC) administration
  Arms: High Dose; Low Dose
Drug: Placebo — SC administration
  Arms: Matching Placebo

SUMMARY:
This study is researching an experimental drug called REGN7544 (called "study drug"). The study is focused on participants with POTS.

The aim of the study is to see how safe, tolerable, and effective the study drug is.

The study is looking at several other research questions, including:

* How the study drug changes heart rate and blood pressure in participants with POTS
* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Is diagnosed with POTS and demonstrates consensus criteria (a), (b), (c) and (d) below during screening:

   1. Increase in HR ≥30 beats per minute (BPM) within 10 minutes of changing from supine to a standing position, as described in the protocol
   2. Absence of orthostatic hypotension, defined as a decrease in systolic blood pressure (SBP) >20 mm Hg within 3 minutes of standing
   3. Absence of other conditions explaining orthostatic tachycardia in the judgment of the investigator, as defined in the protocol
   4. Ongoing episodic symptoms consistent with POTS (for example, lightheadedness, palpitations, tremulousness, generalized weakness, blurred vision, and fatigue) that are worse with standing and are relieved by lying down and which have been present for ≥3 months
2. During screening, a participant must score ≥3 on the Patient Global Impressions of Severity (PGIS)
3. Has a body mass index between 18 and 35 kg/m2, inclusive

Key Exclusion Criteria:

1. History of hypertension or a seated SBP during screening that is >140 mm Hg
2. SBP during active stand (AS) test during screening, either supine or standing, that is >140 mm Hg systolic on ≥2 measurements
3. Increase in HR <20 BPM within 10 minutes of changing from supine to a standing position, as defined in protocol
4. Is judged by the investigator to have significant heart failure, cardiovascular disease, liver disease, or renal disease (ie, estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m2) based on medical history, physical exam, laboratory studies, and/or electrocardiogram (ECG) performed during screening period
5. Is confined to bed more than 50% of waking hours
6. Within 5 days of screening visit has used medications with direct effects on blood volume, BP, or HR (eg, midodrine, droxidopa, octreotide, clonidine, methyldopa, ivabradine, beta-blockers, calcium channel blockers, pyridostigmine, fludrocortisone, desmopressin, stimulants or intravenous (IV) saline)

NOTE: Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate (HR) from supine to standing (DeltaHR) | At Day 8

SECONDARY OUTCOMES:
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Through 90 Days
Severity of TEAEs | Through 90 Days
DeltaHR | At Day 15 and 29
Supine HR | At Day 8, 15, and 29
Standing HR | At Day 8, 15, and 29
Supine blood pressure (BP) | At Day 8, 15, and 29
Standing BP | At Day 8, 15, and 29
Concentrations of REGN7544 in serum | Through 90 Days
Incidence of anti-drug antibodies (ADAs) to REGN7544 | Through 90 Days
Titer of ADAs to REGN7544 | Through 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (18):
- United States (16):
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - North County Neurology Associates, Carlsbad, California
  - Stanford University, Palo Alto, California
  - Southern California Heart Specialists, Pasadena, California
  - Yale University, New Haven, Connecticut
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's MidAmerica Heart Institute, Kansas City, Missouri
  - New York University Langone, New York, New York
  - Columbia University, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: Study Informational Website — https://pinnacle-study.com/en-us/